CLINICAL TRIAL: NCT02657317
Title: Establishing Efficacy of a Functional-Restoration Based CAM Pain Management Program in a Combat-Injured Veterans Population
Brief Title: Establishing Efficacy of a Functional-Restoration Based CAM Pain Management Program in Post-9/11 Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT008422-01 (NIH); HSC20140396 (Other: UTHSCSA)
Record Dates: First submitted 2015-12-17; First posted 2016-01-15 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain; Traumatic Brain Injury; Posttraumatic Stress Disorder; Depression; Opioid Use Disorder
Keywords: chronic pain; pain management; trauma; ptsd; tbi; opioid medication
MeSH Terms: conditions — Chronic Pain; Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Depression; Opioid-Related Disorders; Agnosia; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FORT-A (Experimental): has been labeled "FORT-A." FORT-A is provided on an outpatient basis and includes 12 daily group pain management and physical therapy sessions spanning three weeks. Group interventions are supplemented by individual psychotherapy, biofeedback, and case staffings. CBT sessions were decreased in favor of CAM components. FORT-A participants will receive 270 minutes (4½ hours) of intervention a day for 12 days over 3 weeks.
  Interventions: Behavioral: FORT-A
- VA Treatment As Usual (Active Comparator): Treatment As Usual (TAU) represents usual VA Care based on "as usual" appointments and referrals from VA providers. TAU can include active medical interventions, psychosocial intervention, and other rehabilitation strategies.
  Interventions: Other: VA Treatment as Usual

INTERVENTIONS:
Behavioral: FORT-A — FORT-A is based on a functional restoration paradigm of pain management in which treatment is interdisciplinary and designed to achieve a functional goal (often specified by the patient; e.g., doing more with family, returning to work). FORT-A includes intensive functional rehabilitation, group-based pain management intervention, and individual interventions tailored to the patient's specific needs (e.g., biofeedback for stress, individual psychotherapy for mood or trauma symptoms).
  Other Names: Functional Restoration for Pain
  Arms: FORT-A
Other: VA Treatment as Usual — VA TAU includes referrals for specialty intervention, rehabilitation, and behavioral health intervention within the VA medical system. Some participants may be referred for care outside of the VA system. The South Texas Veterans Health Care System offers a wide range of pain management services.
  Other Names: TAU
  Arms: VA Treatment As Usual

SUMMARY:
This is a research study of an interdisciplinary pain management program for U.S. military veterans who served during the post-9/11 combat eras (e.g., Operations Iraqi Freedom [OIF], Enduring Freedom [OEF], New Dawn [OND]) presenting with chronic musculoskeletal pain related to military service with comorbid depression and/or posttraumatic stress disorder [PTSD] symptoms and/or mild traumatic brain injury. This study will test the efficacy of an interdisciplinary pain program compared to treatment as usual in the Veterans Health Administration on pain-related disability, opioid medication use, and pain coping.

DETAILED DESCRIPTION:
Study Title

Establishing Efficacy of a Functional Restoration-Based Complementary and Alternative Medicine Pain Management Program in a Combat Injured Veterans Population

Objectives

AIM 1: Assess the efficacy of the Functional Orthopedic Rehab Treatment-Amended (FORT-A) Program for improved pain management outcomes in (N=130) polymorbid OEF/OIF/OND Veterans with chronic musculoskeletal pain (CMP) using a 1:1 randomized clinical trial comparing FORT-A to standard Veterans Affairs (VA) care. We will determine the improvement in pain management outcomes attributable to a fully integrated and manualized interdisciplinary pain program (FORT-A) compared to standard VA care.

AIM 2: Assess the efficacy of FORT-A for decreasing the rate of opioid recidivism (using any opioid for 3 or more days in any 30-day period) compared to standard VA care in a sample of OEF/OIF/OND polymorbid Chronic Musculoskeletal Pain (CMP) Veterans discharged off of opioid medication in VA care since the start of the Opioid Safety Initiative (OSI). Unlike the original FORT trial, this research will formally and prospectively track opioid medication use among polymorbid Veterans to sensitively detect changes in chronic opioid therapy attributable to FORT-A versus VA treatment as usual. FORT-A is expected to produce a significantly lower rate of opioid recidivism by imparting numerous strategies to supplant opioid medication as a pain management strategy.

EXPLORATORY AIM 3: The investigators will assess other psychosocial pain coping constructs twice a week and analyze latent changes in FORT-A and VA-treated Veterans to ascertain their role as pain management mediators

Design and Outcomes

This study is a 1:1 block randomized clinical trial comparing the FORT-A program to treatment as usual for polytrauma OEF/OIF/OND Veterans with prior persistent opioid use and chronic musculoskeletal pain who are eligible for treatment through the South Texas Veterans Health Care System (STVHCS). All participants will be offered Physical Therapy services before enrollment and will be enrolled in the study after completing or denying Physical Therapy (up to 12 sessions as recommended by a Polytrauma Rehabilitation Center [PRC] Physical Medicine & Rehabilitation Physician or other VA medical provider). If they have already completed Physical Therapy (PT) before study enrollment, they will not need to do so again. Also, if the Veteran qualifies but refuses VA Physical Therapy, he or she will still be eligible to enroll in this study and will not be asked to complete PT first. Veterans randomized to VA care (treatment as usual) will then meet with PRC and other VA medical providers per usual standards of care (described below). Those randomized to FORT-A will complete the standardized FORT-A Program (described in detail below). All participants will complete a standardized battery of assessments at pre-treatment (Week 0), post-treatment (Week 4/5), 6-month follow-up (Week 30/31) and 12-month follow-up (Week 56/57).

FORT-A: An amended version of the military Functional Orthopedic Rehabilitation Treatment (FORT) program. For FORT-A, Cognitive and Behavioral Therapy (CBT) components of FORT were diminished and replaced with mindfulness and Acceptance and Commitment Therapy (ACT) components. Individual FORT treatment sessions have been altered in FORT-A to focus on PTSD symptom management using an abbreviated, manualized Prolonged Exposure treatment. FORT-A includes:

* 12 sessions (90-minutes each) of manualized group pain management
* 12 sessions (90-minutes each) of group-based functional restoration Physical Therapy
* 6 sessions (75 minutes each) of individual psychotherapy for pain and PTSD
* 6 sessions (30 minutes each) of biofeedback for pain management
* Weekly interdisciplinary case staffings

VA and PRC Care: The STVHCS PRC is the only self-contained Polytrauma Rehab Center in the VA's nationwide Polytrauma System of Care. The PRC is an interdisciplinary treatment center including: interdisciplinary assessment and treatment, case management, mental health support, physical medicine and rehabilitation (PM&R), physical therapy, speech therapy, prosthetists/orthotists, and other integrated specialty services. Though individual treatment plans may vary, most PRC Veterans will complete a course of Physical Therapy and be followed by a PM&R physician for pain and other symptom management. Pain management with PM&R may include medications, injections, and other palliative medical interventions. The PM&R physicians may also make recommendations about physical function, health behaviors, and mobility.

Outcomes will be measured at pre-treatment, post-treatment, 6-month follow-up and one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Demographics for inclusion in this research include both genders, all racial/ethnic groups, and ages 18-72.
2. Present with chronic musculoskeletal pain (CMP) as a primary pain complaint
3. CMP is accompanied by at least moderate disability based on a score of 20% or more on the Oswestry Disability Index;
4. Consistent with NIH Task Force recommendations, "chronic" CMP has been a problem for the Veteran for at least half the days in the last 3 months and was acquired or exacerbated as part of active duty U.S. military service in the Operations Iraqi Freedom (OIF), Enduring Freedom (OEF), or New Dawn (OND) war eras.
5. CMP presents in the context of comorbid psychiatric symptoms of posttraumatic stress disorder (PTSD; based on a score of 25 or more on the PTSD Checklist-Version 5) and/or depression (based on a score of 10 or more on the Beck Depression Inventory-2).
6. Demonstrate prior "chronic" opioid use (defined as using opioid medication for 20 out of every 30 days over three or more months) and discharged off of persistent opioid medications by a VA provider since the onset of the VA Opioid Safety Initiative (2013).
7. Speak and read/understand English well enough to fully participate in the intervention and to reliably complete assessment measures.
8. The Veteran will be eligible to be a PRC patient (i.e., have multiple trauma related physical and psychological injuries; VA, 2013) and be eligible for Physical Therapy referral through the PRC (though the referral for the same service could also come from another VHA provider). All participants will be offered Physical Therapy services before enrollment and will be enrolled after completing or denying Physical Therapy.

Exclusion Criteria:

1. Actively engaged in an intervention or program specifically targeting opioid use (including those using naloxone).
2. Present with active psychosis or suicidal ideation with intent. These symptoms must be stabilized (i.e., maintained at or below moderate intensity for 6 weeks with no acute episodes requiring higher levels of intervention) through a VHA Psychology or Psychiatry referral and confirmed by the mental health provider before the Veteran is eligible to participate.
3. CMP is not related to or exacerbated by military service during the OEF/OIF/OND combat eras.
4. Present with significantly diminished decision-making capacity (e.g., severe cognitive dysfunction related to severe TBI).
5. Pregnant women
6. Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald D McGeary, PhD, Principal Investigator — University of Texas Health Science Center San Antonio; Blessen Eapen, MD, Principal Investigator — South Texas Veterans Health Care System; Cindy A McGeary, PhD, Principal Investigator — University of Texas Health Science Center San Antonio; Carlos Jaramillo, MD, PhD, Principal Investigator — South Texas Veterans Health Care System
Locations (1):
- South Texas Veterans Health Care System, San Antonio, Texas, United States

REFERENCES:
- [Derived] McGeary DD, Jaramillo C, Eapen B, Blount TH, Nabity PS, Moreno J, Pugh MJ, Houle TT, Potter JS, Young-McCaughan S, Peterson AL, Villarreal R, Brackins N, Sikorski Z, Johnson TR, Tapia R, Reed D, Caya CA, Bomer D, Simmonds M, McGeary CA. Mindfulness-Based Interdisciplinary Pain Management Program for Complex Polymorbid Pain in Veterans: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Oct;103(10):1899-1907. doi: 10.1016/j.apmr.2022.06.012. Epub 2022 Aug 6. PMID 35944602

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FORT-A | VA Treatment As Usual
Started | 50 | 53
Completed | 45 | 50
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FORT-A | VA Treatment As Usual | Total
Number analyzed (Participants) | 50 | 53 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (11.0) | 43.7 (9.4) | 43.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 41 | 40 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 16 | 42
  Not Hispanic or Latino | 24 | 37 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 16 | 21
  White | 36 | 28 | 64
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Oswestry Disability Index (ODI)
Description: self-report disability measure. The ODI is a ten-item self report which assesses an individuals perception of limitation in a number of different life domains due to pain. Each item is scored from 0-5 on a numeric rating scale. Scores for each item is summed into a total score and the total is divided by 50 an multiplied by 100 to generate a total score ranging from 0 to 100. This total score represents a % disability score which can be categorized as Minimal (0-20%), Moderate (21-40%), Severe (41-60%), Crippled (61-80%), or Bed Bound/Exaggerating (81-100%).
Time Frame: Pre-Treatment, Post-Treatment 3 weeks after Pre-Treatment, Follow-Up 6 Months After Post-Treatment, Follow-Up 12 Months After Post-Treatment
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | FORT-A | VA Treatment As Usual
Number analyzed (Participants) | 50 | 53
score on a scale
  Pre-Treatment | 48.6 [42.4 to 54.8] | 45.1 [39.5 to 50.7]
  Post-Treatment | 38.3 [33.5 to 43.1] | 47.8 [42.5 to 53.0]
  6-Month Follow-up | 37.6 [32.7 to 42.5] | 47.1 [41.7 to 52.5]
  12-Month Follow-up | 37.9 [33.0 to 42.7] | 45.7 [40.1 to 51.2]
Statistical Analysis 1: Comparison: FORT-A vs VA Treatment As Usual; To detect a medium effect (d = 0.50) at 2-sided α = 0.05, 50 participants were needed in each study arm (total N = 100). We anticipated 30% attrition in each arm. Data for the primary aim were analyzed using generalized linear mixed models adjusting for baseline levels of prognostic variable and using random intercepts at the level of participants. The primary analysis was based on intent-to-treat; Test type: Superiority; p = .001, GLMM; Mean Difference (Final Values) = -9.1, 95% CI 2-sided [-14.4 to -3.7]

ADVERSE EVENTS:
Time Frame: 1 year
Description: definitions consistent with clinicaltrials.gov definitions
Arm/Group | FORT-A | VA Treatment As Usual
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/53
Other Adverse Events (participants affected / at risk) | 15/50 | 13/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FORT-A (N=50) | VA Treatment As Usual (N=53)
Knee Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (10) — Pain in knee
Increased Anxiety (Nervous system disorders) | 2 (4) | 8 (9)
Increased Nightmares (Psychiatric disorders) | 2 (2) | 0 (0) — Subject experience more nightmares than usual
Increased Anger (Psychiatric disorders) | 3 (3) | 0 (0)
Pain in right let (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 12 (14)
Numbness and tingling in feet (Nervous system disorders) | 2 (2) | 2 (2)
Cold and numbness in feet (Nervous system disorders) | 1 (1) | 0 (0)
Neck discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) — Pressure at back of neck
General pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Sleep difficulties due to discontinued opioid (Nervous system disorders) | 1 (1) | 0 (0)
Increase in pain due to discontinuation of opioid (General disorders) | 2 (2) | 2 (2)
Increased irritability due to discontinuation of opioids (Psychiatric disorders) | 1 (1) | 1 (1)
Increase in headaches due to discontinuation of opioids (Nervous system disorders) | 1 (1) | 0 (0)
Whole body aches (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 10 (11) — new dull pain in mid back possibly due to going swimming

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02657317/Prot_SAP_000.pdf